CLINICAL TRIAL: NCT04699747
Title: Investigating the Utility of Demyelination Tracer [18F]3F4AP in Controls and Multiple Sclerosis Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Brugarolas, Assistant Professor of Radiology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P002459
Record Dates: First submitted 2020-12-16; First posted 2021-01-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Demyelination; Brain imaging; Positron Emission Tomography; Radiopharmaceutical
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Intervention Model Description: Drug: F-18 3F4AP PET scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple sclerosis (Experimental): F-18 3F4AP PET Scan
  Interventions: Drug: F-18 3F4AP
- Healthy controls (Active Comparator): F-18 3F4AP PET Scan
  Interventions: Drug: F-18 3F4AP

INTERVENTIONS:
Drug: F-18 3F4AP — Subjects will be injected once per imaging session (a maximum of 2 imaging sessions) with up to 10 mCi (±20%) of 18-F 3F4AP as a rapid intravenous bolus (within 1 min).
  Other Names: [18F]3F4AP

SUMMARY:
Our overall objective is to obtain an initial assessment of the potential value of using [18F]3F4AP for imaging demyelinating diseases such as multiple sclerosis:

* Aim 1) Assess the safety of [18F]3F4AP in healthy volunteers and subjects with multiple sclerosis (MS). Hypothesis 1: Administration of [18F]3F4AP will result in no changes in vitals or other adverse events.
* Aim 2) Assess the pharmacokinetics of a bolus infusion of [18F]3F4AP in humans including healthy volunteers and MS patients. Hypothesis 2: the pharmacokinetics of [18F]3F4AP at the whole brain level will be similar in controls and MS subjects. The kinetics in demyelinated lesions will be slower than in healthy control areas.
* Aim 3) Assess the reproducibility of [18F]3F4AP in humans. Hypothesis 3: the test/retest variability of [18F]3F4AP within the same subject will be lower than 10%.
* Aim 4) Correlate MR brain images with [18F]3F4AP PET brain images. Hypothesis 4A: all the lesions seen on the MRI will show increased signal (VT or SUV) on the PET images. Hypothesis 4B: some of the lesions on the MRI will show increased signal (VT or SUV) on the PET but not all.
* Aim 5) Correlate [18F]3F4AP PET signal with neuropsychological testing in people with MS. Hypothesis 5: increased PET signal (VT or SUV) will correlate with impaired Single Digit Modality Test (SDMT) scores.
* Aim 6) Correlate [18F]3F4AP PET signal with EDSS score in people with MS. Hypothesis 6: increased PET signal (VT or SUV) will correlate with higher EDSS scores.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 and <65 years of age;
* Able to understand and provide informed consent prior to study procedures

Exclusion Criteria:

* Subjects with known structural brain disease (e.g. brain tumor or stroke);
* Any contraindication to MRI and/or PET, including:

  * Subjects with life vest;
  * Subjects with implanted heart device (e.g. ICD, Pacemaker);
  * Subjects with metallic fragment or foreign body;
  * Subjects with other form of devices or prosthesis that are not MRI compatible, such as insulin pump, joint replacement, hearing aid, cochlear implant, permanent contraceptive devices, etc.;
  * Subjects with severe claustrophobia
  * Relative or absolute contraindication to Dotarem contrast:
* history of renal disease including acute or chronic severe renal insufficiency (glomerular filtration rate <60 mL/min/1.73m2);
* history of diabetes mellitus, systemic lupus, multiple myeloma, nephrogenic systemic fibrosis, and other co-morbidities;
* History of hypersensitive reactions to Dotarem and/or gadolinium contrast agent;
* Radiation exposure exceeds current Radiology Department guidelines (i.e., 50 mSv in the prior 12 months);
* Female subjects only: Positive serum pregnancy test, or lactating, or possibility of pregnancy cannot be ruled out prior to dosing;
* Inability to provide written informed consent;
* Any clinically significant acute or unstable physical or psychiatric condition, judged by the investigators based on medical history or screening physical examination, to be incompatible with the study;
* Any physical or psychiatric condition judged by the investigators to be incompatible with the study, based on medical history or screening physical examination;
* Abnormal results on blood tests judged by the investigators to be incompatible with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Binding of 18-F 3F4AP in the brain of healthy volunteers and multiple sclerosis subjects | Baseline
  Binding of the tracer will be quantified using volumes of distribution (VTs). Volume of distribution is the ratio of tracer concentration in tissue to plasma at equilibrium and will be determined using standard pharmacokinetic methods (Innis et al, J Cereb Blood Flow Metab. 2007; 27(9): 1533-1539).
Number of participants with adverse events related to tracer administration as assessed by CTCAE v4.0 | 5 years
  Determine number of participants adverse events related to tracer administration as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Binding of 18-F 3F4AP in brain lesions of multiple sclerosis subjects | Baseline
  Binding of the tracer in the lesions will be quantified using volumes of distribution (VTs). Lesions will be delineated based on 3D FLAIR MRI using standardized methods.
Within-subject variability in healthy controls and multiple sclerosis subjects | Retest within 3 months of baseline
  Within-subject variability (test/retest variability or TRV) of the VT in healthy volunteers and multiple sclerosis subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiss A, Michaelson NM, Russo AW, Ramos-Torres KM, Sun Y, DaSilva NE, Noel JM, Liu F, Gong K, Huang SY, Popko B, Baker S, Klawiter EC, Brugarolas P. First evaluation in multiple sclerosis using PET tracer [18F]3F4AP demonstrates heterogeneous binding across lesions. Eur J Nucl Med Mol Imaging. 2026 Jan;53(2):1125-1138. doi: 10.1007/s00259-025-07454-1. Epub 2025 Aug 5. PMID 40759830